CLINICAL TRIAL: NCT06632561
Title: Benefits of Empagliflozin in Patients With Heart Failure and Reduced Ejection Fraction Without Diabetes Mellitus
Acronym: HFrEF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ashraf Wasfy Beshay Aziz (Other)
Responsible Party: Sponsor-Investigator, Ashraf Wasfy Beshay Aziz, Cardiology Specialist, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/06072021/Aziz
Record Dates: First submitted 2024-10-06; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin arm (Experimental): 37 patients received Empagliflozin 10 mg/day in addition to their guideline-directed medical therapy for HF
  Interventions: Drug: Empagliflozin 10 mg
- Placebo arm (Placebo Comparator): 37 patients received placebo in addition to their guideline-directed medical therapy for HF
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 mg — Empagliflozin (a sodium-glucose cotransporter-2 inhibitor) 10 mg one tablet daily dose for 6 months
  Arms: Empagliflozin arm
Drug: Placebo — Sugar pills one tablet daily for 6 months
  Arms: Placebo arm

SUMMARY:
The study is a short to mid-term randomized single-blind placebo controlled study that aimed to detect the effects of empagliflozin (a sodium-glucose cotransporter-2 inhibitor) compared to placebo on LV end-diastolic and end-systolic volumes, LV ejection fraction, N-terminal pro-B-type natriuretic peptide (NT-proBNP), functional capacity and quality of life (QoL) among non-diabetic patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory non-diabetic adult male and non-pregnant female patients with established diagnosis of heart failure (HF) New York Heart Association functional class II-IV and left ventricular ejection fraction (LVEF) ≤ 40% (calculated by echocardiography within the previous 6 months before randomization).
* Patients should have stable symptoms and stable guideline-directed medical therapy for HF within the last 3 months before randomization. It was mandatory that all patients have reached the maximum tolerated doses of guideline-directed medical therapy for HF and are regular on them for at least 3 months before participation.
* Patients were not known to be diabetic and have no history of diabetes remission and their baseline glycosylated hemoglobin (HbA1c) should have been < 5.7%.
* Patients have never been on SGLT2 inhibitor therapy before.
* Estimated glomerular filtration rate (eGFR) should have been ≥ 45 mL/min/1.73 m² using the chronic kidney disease Epidemiology Collaboration (CKD-EPI) creatinine equation (2009)

Exclusion Criteria:

* Women who were pregnant at time of selection, possibly pregnant, breast-feeding, or planning to become pregnant during the study period.
* Patients who had acute coronary syndrome, cardiac surgery, stroke or transient ischemic attack (TIA) within the last 3 months before randomization.
* Patients who had infiltrative cardiomyopathy, muscular dystrophies, hypertrophic cardiomyopathy, peripartum cardiomyopathy, pericardial restriction or chemotherapy induced cardiomyopathy within 12 months before randomization.
* Patients with severe valvular heart disease.
* Patients who had acute decompensated HF or were on continuous parenteral inotropic agents with 3 months before randomization.
* Patients who had cardiac resynchronization therapy (CRT) implantation within 3 months before randomization.
* History of recurrent urinary tract infection, cancer or any life threatening condition or psychiatric disease incompatible with being in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
The changes in LV volumes (mL) | From enrollment to the end of treatment at 6 months
  To measure the changes in of Left Ventricular end-diastolic volume (LVEDV) (mL) and Left Ventricular end-systolic volume (LVESV) (mL) via transthoracic echocardiography using the modified Simpson's rule (the biplane disk summation approach).
  Then the change from baseline to the 6th month was compared within each group separately and the means of variables were compared between both groups.
The changes in of Left Ventricular Ejection Fraction (LVEF) (%) | From enrollment to the end of treatment at 6 months
  To measure the changes in of Left Ventricular Ejection Fraction (LVEF) (%) via transthoracic echocardiography using the modified Simpson's rule (the biplane disk summation approach).
  Then the change from baseline to the 6th month was compared within each group separately and the means of variables were compared between both groups.

SECONDARY OUTCOMES:
The changes in the N-terminal pro-B-type natriuretic peptide (NT-proBNP) (pg/mL) | From enrollment to the end of treatment at 6 months
  Measurement of N-terminal pro-B-type natriuretic peptide (NT-proBNP) (pg/mL) at baseline and at the end of treatment phase after 6 months within both study arms via the electrochemiluminescence immunoassay "ECLIA".
  Then the change from baseline to the 6th month was compared within each group separately and the means of variables were compared between both groups.
The changes in 6 minute walk test (meters) | From enrollment to the end of treatment at 6 months
  Measurement of 6 minute walk test (meters) at baseline and at the end of treatment phase after 6 months within both study arms.
  Then the change from baseline to the 6th month was compared within each group separately and the means of variables were compared between both groups.
The changes in the Minnesota Living with Heart Failure Questionnaire (MLHFQ) (points) | From enrollment to the end of treatment at 6 months
  Measurement of the Minnesota Living with Heart Failure Questionnaire (MLHFQ) (points) at baseline and at the end of treatment phase after 6 months within both study arms.
  Then the change from baseline to the 6th month was compared within each group separately and the means of variables were compared between both groups.

OTHER OUTCOMES:
a (five points or more) improvement in the Minnesota Living with Heart Failure Questionnaire | From enrollment to the end of treatment at 6 months
  Since a five point change in MLHFQ is considered clinically meaningful, we have performed an exploratory analysis to compare the proportion of patients with ≥5 points improvement in MLHFQ in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham B Mahmoud, Professor of Cardiology, Study Chair — Beni-Suef University; Mohammad Sh Awad, Assistant Professor Cardiology, Study Director — Beni-Suef University; Mohammed M Tohamy, Lecturer of Cardiology, Study Director — Beni-Suef University
Locations (1):
- Beni-Suef University, BeniSuef, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Santos-Gallego CG, Vargas-Delgado AP, Requena-Ibanez JA, Garcia-Ropero A, Mancini D, Pinney S, Macaluso F, Sartori S, Roque M, Sabatel-Perez F, Rodriguez-Cordero A, Zafar MU, Fergus I, Atallah-Lajam F, Contreras JP, Varley C, Moreno PR, Abascal VM, Lala A, Tamler R, Sanz J, Fuster V, Badimon JJ; EMPA-TROPISM (ATRU-4) Investigators. Randomized Trial of Empagliflozin in Nondiabetic Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2021 Jan 26;77(3):243-255. doi: 10.1016/j.jacc.2020.11.008. Epub 2020 Nov 13. PMID 33197559